CLINICAL TRIAL: NCT00196742
Title: Fabry Disease Registry Protocol
Brief Title: Fabry Disease Registry & Pregnancy Sub-registry
Status: Recruiting | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DIREGC07006; AGAL19211 (Other: Genzyme, a Sanofi cmpany); U1111-1294-8298 (Registry Identifier: ICTRP)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Fabry Disease
Keywords: alpha Galactosidase A; aGAL (alpha-galactosidase); Fabry; GL3 (globotriaosylceramide); Anderson-Fabry Disease; angiokeratomas; GLA deficiency (gene deficiency); errors in metabolism
MeSH Terms: conditions — Fabry Disease; Angiokeratoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Fabry disease: No experimental intervention is given. A patient with Fabry Disease will undergo clinical assessments and receive standard of care treatment as determined by the patient's physician.
- Pregnant women with confirmed diagnosis of Fabry: No experimental intervention is given. Pregnant women with confirmed diagnosis of Fabry that are participating in the Fabry Registry and consented to participate in the Fabry Sub-registry, regardless of whether she is receiving disease-specific therapy (such as ERT with agalsidase beta) and irrespective of the commercial product with which she may be treated.

SUMMARY:
The Fabry Registry is an ongoing, international multi-center, strictly observational program that tracks the routine clinical outcomes for patients with Fabry disease, irrespective of treatment status. No experimental intervention is involved; patients in the Registry undergo clinical assessments and receive care as determined by the patient's treating physician.

The primary objectives of the Registry are:

* To enhance the understanding of the variability, progression, and natural history of Fabry disease, including heterozygous females with the disease;
* To assist the Fabry medical community with the development of recommendations for monitoring patients and reports on patient outcomes to help optimize patient care;
* To characterize and describe the Fabry population as a whole;
* To evaluate the long-term safety and effectiveness of Fabrazyme®

Fabry Pregnancy Sub-registry: This Sub-registry is a multicenter, international, longitudinal, observational, and voluntary program designed to track pregnancy outcomes for any pregnant woman enrolled in the Fabry Registry, regardless of whether she is receiving disease-specific therapy (such as enzyme replacement therapy with agalsidase beta) and irrespective of the commercial product with which she may be treated. Data from the Sub-registry are also used to fulfill various global regulatory requirements, to support product development/reimbursement, and for other research and non-research-related purposes. No experimental intervention is given; thus a patient will undergo clinical assessments and receive standard of care treatment as determined by the patient's physician. If a patient consents to this Sub-registry, information about the patient's medical and obstetric history, pregnancy, and birth will be collected, and, if a patient consents to data collection for her infant, data on infant growth through month 36 postpartum will be collected.

ELIGIBILITY:
Inclusion Criteria

* Fabry Registry: All patients with a confirmed diagnosis of Fabry disease who have signed the informed consent and patient authorization form(s) are eligible for inclusion. Confirmed diagnosis is defined as a documented deficiency in plasma or leukocyte αGAL (alpha-galactosidase) enzyme activity and/or mutation(s) in the gene coding for αGAL.
* Fabry Pregnancy Sub-registry:

  * Eligible women must:

    * be enrolled in the Fabry Registry.
    * be pregnant, or have been pregnant with appropriate medical documentation available.
    * provide a signed informed consent and authorization form(s) to participate in the Sub-Registry prior to any Sub-Registry-related data collection being performed.

Exclusion Criteria Fabry Registry: There are no exclusion criteria. Fabry Pregnancy Sub-registry: There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a confirmed diagnosis of Fabry disease are eligible for inclusion in the Registry.
  For Fabry Pregnancy Sub-registry: It is recommended that pregnancy data be collected on eligible women regardless of infant enrollment. In the event of patients having multiple pregnancies, data collection for each individual pregnancy is encouraged for all women enrolled in this Sub-Registry.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2001-07-31 (Actual); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Fabry Registry: To evaluate the long-term safety and effectiveness of Fabrazyme® | 33 years
  The primary purpose of this Registry is to describe the development and progression of Fabry disease in a representative global population. As Fabry is not a well-described disease this longitudinal program has a wide variety of "primary" outcomes including antibody testing as well as complication outcomes (eg, QoL, cognitive testing) which are measured over time. Additionally, as it is subject to what is collected by clinical sites at the time of visit it is unknown the amount of data that will be available for analyses.
Fabry Pregnancy Sub-registry: pregnancy outcomes, including complications and infant growth | 33 years
  The primary objective of this Sub-registry is to track pregnancy outcomes, including complications and infant growth, in all women with Fabry disease during pregnancy, regardless of whether they receive disease-specific therapy, such as ERT with agalsidase beta.
  This Sub-registry augments the routine monitoring and data collection recommended by the Fabry Registry. The Sub-registry aims to collect patient assessments from the ante- and perinatal periods and postpartum follow-up. Neonatal assessments and periodic pediatric assessments will also be collected.

SECONDARY OUTCOMES:
Fabry Register: Monitor factors associated with the efficacy of Fabry disease treatments | 33 years
  A secondary endpoint is to monitor those factors associated with the efficacy of Fabry disease treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Genzyme, a Sanofi Company
Locations (281):
- United States (92):
  - University of Alabama Birmingham- Nephrology- Site Number : 840018, Birmingham, Alabama
  - University of Alabama Birmingham- Nephrology- Site Number : 840073, Birmingham, Alabama
  - Phoenix Children's Hospital- Site Number : 840003, Phoenix, Arizona
  - University of Arizona- Site Number : 840015, Tucson, Arizona
  - Arkansas Childrens Hospital- Site Number : 840109, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences- Site Number : 840113, Little Rock, Arkansas
  - University of California at Irvine- Site Number : 840036, Irvine, California
  - Southern California Permanente Medical Group- Site Number : 840108, Los Angeles, California
  - USC Health Sciences Center Dept of Genetics- Site Number : 840082, Los Angeles, California
  - UCLA School Of Medicine- Site Number : 840088, Los Angeles, California
  - Children's Hospital Oakland- Site Number : 840029, Oakland, California
  - Children's Hospital of Orange County- Site Number : 840074, Orange, California
  - Stanford Unviersity MC Dept of Genetics- Site Number : 840022, Palo Alto, California
  - UC Davis MIND Institute- Site Number : 840010, Sacramento, California
  - Kaiser Permanente Hospital- Site Number : 840042, Sacramento, California
  - University of California at San Diego- Site Number : 840007, San Diego, California
  - University of California at San Francisco- Site Number : 840051, San Francisco, California
  - Yale - Site Number : 840047, New Haven, Connecticut
  - Children's National Medical Center- Site Number : 840067, Washington D.C., District of Columbia
  - University Hematology Oncology- Site Number : 840075, Coral Springs, Florida
  - University of Florida Dept of Genetics- Site Number : 840083, Gainesville, Florida
  - University of Florida Pediatrics Genetics- Site Number : 840121, Jacksonville, Florida
  - University Of Miami SOM- Site Number : 840006, Miami, Florida
  - University of Florida-Genetics- Site Number : 840096, Tampa, Florida
  - Emory University School of Medicine- Human Genetics- Site Number : 840060, Decatur, Georgia
  - University of Colorado at Denver Genetics- Site Number : 840068, Aurora, Illinois
  - Ann and Robert Lurie Children's Hospital- Site Number : 840013, Chicago, Illinois
  - Rush University Medical Center Genetics- Site Number : 840079, Chicago, Illinois
  - Indianapolis University School of Medicine- Site Number : 840027, Indianapolis, Indiana
  - University of Iowa- Site Number : 840032, Iowa City, Iowa
  - University of Kansas Medical Center- Site Number : 840071, Kansas City, Kansas
  - University of Louisville- Genetics- Site Number : 840030, Louisville, Kentucky
  - Ochsner Medical Center- Site Number : 840120, Baton Rouge, Louisiana
  - Tulane University Medical Center- Site Number : 840001, New Orleans, Louisiana
  - Maine Medical Center Pediatrics- Site Number : 840064, Portland, Maine
  - John Hopkins- Site Number : 840044, Baltimore, Maryland
  - Massachusetts General Hospital-Genetics- Site Number : 840062, Boston, Massachusetts
  - Boston Children's Hospital - PIN- Site Number : 840092, Boston, Massachusetts
  - Brigham and Women's Hospital-Neurology- Site Number : 840103, Boston, Massachusetts
  - Baystate Health- Site Number : 840002, Springfield, Massachusetts
  - University of Michigan Pediatrics- Site Number : 840107, Ann Arbor, Michigan
  - Children's Hospital of Michigan- Site Number : 840066, Detroit, Michigan
  - Spectrum for Health- Site Number : 840019, Grand Rapids, Michigan
  - Infusion Associates- Site Number : 840050, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota- Site Number : 840046, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota- Site Number : 840114, Minneapolis, Minnesota
  - University of Minnesota Medical Center Pediatrics- Site Number : 840076, Minneapolis, Minnesota
  - University of Missouri Health System Department of Genetics- Site Number : 840031, Columbia, Missouri
  - Washington University of St. Louis- Site Number : 840100, St Louis, Missouri
  - Shodair Children's Hospital- Site Number : 840090, Helena, Montana
  - University of Nebraska Medical Center- Pediatrics- Site Number : 840084, Omaha, Nebraska
  - Children's Specialty Center of Nevada- Site Number : 840008, Las Vegas, Nevada
  - Cooper Health Center- Site Number : 840098, Camden, New Jersey
  - Joseph M. Sanzari Children's Hospital- Site Number : 840101, Hackensack, New Jersey
  - Atlantic Health System- Site Number : 840099, Morristown, New Jersey
  - St. Peter's University Hospital- Site Number : 840016, New Brunswick, New Jersey
  - St. Joseph's Children's Hospital- Site Number : 840057, Paterson, New Jersey
  - Northwell Health- Site Number : 840102, Manhasset, New York
  - New York University School Of Medicine- Site Number : 840040, New York, New York
  - Metropolitan Hospital Center- Site Number : 840110, New York, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 840080, New York, New York
  - University of Rochester Medical Center SOM- Site Number : 840105, Rochester, New York
  - State University of New York- Site Number : 840052, Syracuse, New York
  - New York Medical College- Site Number : 840039, Valhalla, New York
  - Carolinas Medical Center- Site Number : 840065, Charlotte, North Carolina
  - Duke University Medical Center Genetics Dept- Site Number : 840045, Durham, North Carolina
  - Cincinnati Children's Hospital-Genetics- Site Number : 840033, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 840119, Cleveland, Ohio
  - Cleveland Clinic Foundation Pediatrics- Site Number : 840048, Cleveland, Ohio
  - Nationwide Children's Hospital - PIN- Site Number : 840091, Columbus, Ohio
  - Ohio State University Department of Genetics- Site Number : 840097, Columbus, Ohio
  - LSD Data Registry Site LLC- Site Number : 840094, Dublin, Ohio
  - Oregon Health & Science University (OHSU)- Site Number : 840116, Portland, Oregon
  - Oregon Health and Scinece University- Site Number : 840038, Portland, Oregon
  - Geisinger- Site Number : 840111, Danville, Pennsylvania
  - Penn State University Medical Center-Neurology- Site Number : 840104, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia HUP Medical Genetics- Site Number : 840089, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia- Site Number : 840034, Philadelphia, Pennsylvania
  - University of Pittsburgh- Site Number : 840023, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Genetics- Site Number : 840053, Providence, Rhode Island
  - Greenwood Genetcs- Site Number : 840055, Greenville, South Carolina
  - Vanderbilt University Hospital-Pediatrics- Site Number : 840049, Nashville, Tennessee
  - Baylor Research Center- Site Number : 840058, Dallas, Texas
  - Cook Children's Health Care System- Site Number : 840024, Fort Worth, Texas
  - University of Utah Department of Medical Genetics- Site Number : 840043, Salt Lake City, Utah
  - University of Virginia School of Medicine-Pediatrics- Site Number : 840078, Charlottesville, Virginia
  - O&O Alpan, LLC- Site Number : 840025, Fairfax, Virginia
  - Children's Hospital of the Kings Daughters- Site Number : 840072, Norfolk, Virginia
  - Seattle Children's Hospital- Site Number : 840028, Seattle, Washington
  - University Of Washington Medical Center- Site Number : 840059, Seattle, Washington
  - Mary Bridge Children's Outpatient Center- Site Number : 840115, Tacoma, Washington
  - Children's Hospital of Wisconsin-Pediatrics- Site Number : 840054, Milwaukee, Wisconsin
- Argentina (10):
  - Investigational Site Number : 153280, Berazategui, Buenos Aires
  - Investigational Site Number : 153260, Caba, Buenos Aires, Buenos Aires
  - Investigational Site Number : 153032, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Investigational Site Number : 153250, San Isidro, Buenos Aires, Buenos Aires
  - Investigational Site Number : 153194, Catamarca, Catamarca Province
  - Investigational Site Number : 153172, Buenos Aires
  - Investigational Site Number : 153130, Buenos Aires
  - Investigational Site Number : 032005, La Rioja
  - Investigational Site Number : 153270, La Rioja Province
  - Investigational Site Number : 032004, Santa Fe
- Australia (6):
  - Investigational Site Number : 036013, Westmead, New South Wales
  - Investigational Site Number : 151069, Westmead, New South Wales
  - Investigational Site Number : 153063, Brisbane, Queensland
  - Investigational Site Number : 151002, Adelaide, South Australia
  - Investigational Site Number : 153040, Parkville, Victoria
  - Investigational Site Number : 153090, Perth, Western Australia
- Belgium (8):
  - Investigational Site Number : 150722, Antwerp
  - Investigational Site Number : 153133, Antwerp
  - Investigational Site Number : 153001, Brussels
  - Investigational Site Number : 0560008, Brussels
  - Investigational Site Number : 150517, Brussels
  - Investigational Site Number : 151668, Leuven
  - Investigational Site Number : 154275, Liège
  - Investigational Site Number : 153100, Seraing
- Brazil (11):
  - Clínica Senhor do Bonfim LTDA- Site Number : 076008, Feira de Santana, Estado de Bahia
  - Medicordis- Site Number : 076009, Brasília, Federal District
  - Hospital Geral e Maternidade de Cuiabá- Site Number : 076006, Cuiabá, Mato Grosso
  - CTDR - Centro de Tratamento de Doenças Renais EIRELI- Site Number : 076007, Uberlândia, Minas Gerais
  - Instituto do Rim do Paraná- Site Number : 076004, Curitiba, Paraná
  - Instituto de Medicina Integral Professor Fernando Figueira - IMIP - Site Number : 076005, Recife, Pernambuco
  - Saúde Center Clínica - Clínica Médica Nossa Senhora de Fátima - Site Number : 076002, Tapejara, Rio Grande do Sul
  - Hospital Universitário Professor Polydoro Ernani de São Thiago - UFSC- Site Number : 076012, Florianópolis, Santa Catarina
  - Hospital e Maternidade Celso Pierro - PUC-Campinas- Site Number : 076013, Campinas, São Paulo
  - Serviço de Terapia Renal de Ourinhos- Site Number : 076011, Ourinhos, São Paulo
  - Instituto de Genética e Erros Inatos do Metabolismo- Site Number : 076001, São Paulo
- Bulgaria (2):
  - Investigational Site Number : 153169, Sofia
  - Investigational Site Number : 100001, Sofia
- Canada (14):
  - Investigational Site Number : 124014, Calgary, Alberta
  - Investigational Site Number : 124002, Edmonton, Alberta
  - Investigational Site Number : 124010, Vancouver, British Columbia
  - Investigational Site Number : 124011, Vancouver, British Columbia
  - Investigational Site Number : 124019, Winnipeg, Manitoba
  - Investigational Site Number : 124022, Moncton, New Brunswick
  - Investigational Site Number : 124023, St. John's, Newfoundland and Labrador
  - Investigational Site Number : 124008, Halifax, Nova Scotia
  - Investigational Site Number : 124005, Kingston, Ontario
  - Investigational Site Number : 124021, London, Ontario
  - Investigational Site Number : 124006, Toronto, Ontario
  - Investigational Site Number : 124009, Toronto, Ontario
  - Investigational Site Number : 124013, Montreal, Quebec
  - Investigational Site Number : 124001, Sherbrooke, Quebec
- Chile (5):
  - Investigational Site Number : 152004, Antofagasta
  - Investigational Site Number : 152001, Coquimbo
  - Investigational Site Number : 152003, Iquique
  - Investigational Site Number : 152002, Santiago
  - Investigational Site Number : 152005, Vallenar
- China (6):
  - Investigational Site Number : 153165, Beijing
  - Investigational Site Number : 1560003, Hangzhou
  - Investigational Site Number : 1560002, Jinan
  - Investigational Site Number : 1560004, Nanjing
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 153163, Shanghai
- Investigational Site Number : 170001, Bogotá, Colombia
- Croatia (2):
  - Investigational Site Number : 1910001, Rijeka
  - Investigational Site Number : 1910002, Zagreb
- Investigational Site Number : 153126, Prague, Czechia
- Denmark (2):
  - Investigational Site Number : 153041, Copenhagen
  - Investigational Site Number : 151229, København Ø
- Investigational Site Number : 153106, Tartu, Estonia
- Investigational Site Number : 153024, Turku, Finland
- France (6):
  - Investigational Site Number : 250005, Bordeaux
  - Investigational Site Number : 250002, Bron
  - Investigational Site Number : 250001, Garches
  - Investigational Site Number : 250007, Lille
  - Investigational Site Number : 250004, Saint-Priest-en-Jarez
  - Investigational Site Number : 250009, Strasbourg
- Germany (4):
  - Investigational Site Number : 153013, Berlin
  - Investigational Site Number : 154150, Giessen
  - Investigational Site Number : 153147, Münster
  - Investigational Site Number : 153011, Würzburg
- Investigational Site Number : 344001, Kowloon, Hong Kong
- Hungary (4):
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480003, Létavértes
  - Investigational Site Number : 3480005, Pécs
  - Investigational Site Number : 3480004, Sopron
- India (4):
  - Investigational Site Number : 356003, Ahmedabad
  - Investigational Site Number : 356001, Kolkata
  - Investigational Site Number : 3560004, Secunderabad
  - Investigational Site Number : 356002, Vellore
- Investigational Site Number : 360001, Jakarta, Indonesia
- Italy (15):
  - Investigational Site Number : 380002, Bassano del Grappa
  - Investigational Site Number : 380019, Bologna
  - Investigational Site Number : 380004, Florence
  - Investigational Site Number : 380013, Florence
  - Investigational Site Number : 380005, Genova
  - Investigational Site Number : 380009, Milan
  - Investigational Site Number : 380006, Milan
  - Investigational Site Number : 380003, Modena
  - Investigational Site Number : 380010, Monza
  - Investigational Site Number : 380008, Napoli
  - Investigational Site Number : 380007, Rimini
  - Investigational Site Number : 380012, Roma
  - Investigational Site Number : 380011, Torino
  - Investigational Site Number : 380001, Udine
  - Investigational Site Number : 380014, Vittoria
- Japan (6):
  - Investigational Site Number : 392007, Kobe, Hyōgo
  - Investigational Site Number : 153201, Nangoku-shi, Kochi
  - Investigational Site Number : 153205, Abeno-ku, Osaka
  - Investigational Site Number : 153217, Chiba
  - Investigational Site Number : 392006, Niigata
  - Investigational Site Number : 153204, Tokyo
- Lithuania (2):
  - Investigational Site Number : 154244, Vilnius
  - Investigational Site Number : 154652, Vilnius
- Malaysia (2):
  - Investigational Site Number : 458002, Kuala Lumpur
  - Investigational Site Number : 458001, Kuala Pahang
- Netherlands (2):
  - Investigational Site Number : 151171, Amsterdam
  - Investigational Site Number : 153004, Amsterdam
- Investigational Site Number : 153141, Bergen, Norway
- Investigational Site Number : 604002, Callao, Peru
- Investigational Site Number : 608001, Manila, Philippines
- Investigational Site Number : 150575, Warsaw, Poland
- Portugal (2):
  - Investigational Site Number : 620005, Lisbon
  - Investigational Site Number : 620001, Porto
- Romania (3):
  - Investigational Site Number : 154099, Bucharest
  - Investigational Site Number : 154164, Bucharest
  - Investigational Site Number : 153081, Cluj-Napoca
- Russia (3):
  - Investigational Site Number : 643001, Moscow
  - Investigational Site Number : 643003, Nizhny Novgorod
  - Investigational Site Number : 643002, Saint-Peterburg
- Investigational Site Number : 682002, Al Mubarraz, Saudi Arabia
- Investigational Site Number : 6880001, Novi Sad, Serbia
- Investigational Site Number : 702001, Singapore, Singapore
- Investigational Site Number : 703001, Bratislava, Slovakia
- Investigational Site Number : 705001, Slovenj Gradec, Slovenia
- South Korea (14):
  - Investigational Site Number : 153178, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 154208, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 157176, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 153180, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 153196, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 154246, Busan
  - Investigational Site Number : 153191, Daejeon
  - Investigational Site Number : 153228, Jeju City
  - Investigational Site Number : 153192, Seoul
  - Investigational Site Number : 151149, Seoul
  - Investigational Site Number : 153188, Seoul
  - Investigational Site Number : 153212, Seoul
  - Investigational Site Number : 153222, Seoul
  - Investigational Site Number : 154273, Suwon
- Spain (11):
  - Investigational Site Number : 154146, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 154159, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 153237, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 154147, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 154135, Barakaldo, Basque Country
  - Investigational Site Number : 154204, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 153213, Vigo, Pontevedra [Pontevedra]
  - Investigational Site Number : 154136, Tarragona, Tarragona [Tarragona]
  - Investigational Site Number : 153067, Barcelona
  - Investigational Site Number : 153077, Barcelona
  - Investigational Site Number : 154123, Barcelona
- Sweden (2):
  - Investigational Site Number : 153050, Gothenburg
  - Investigational Site Number : 151484, Stockholm
- Taiwan (15):
  - Investigational Site Number : 151500, Chiayi City
  - Investigational Site Number : 154093, Chiayi City
  - Investigational Site Number : 152152, Hualien City
  - Investigational Site Number : 152244, Kaohsiung City
  - Investigational Site Number : 153088, Kaohsiung City
  - Investigational Site Number : 152246, Kaohsiung City
  - Investigational Site Number : 151534, New Taipei City
  - Investigational Site Number : 151179, Taichung
  - Investigational Site Number : 151181, Taichung
  - Investigational Site Number : 153248, Tainan
  - Investigational Site Number : 152153, Tainan
  - Investigational Site Number : 151182, Taipei
  - Investigational Site Number : 152321, Taipei
  - Investigational Site Number : 152226, Taipei
  - Investigational Site Number : 153158, Tao Yuan County
- Thailand (4):
  - Investigational Site Number : 764003, Bangkok
  - Investigational Site Number : 764004, Bangkok
  - Investigational Site Number : 764001, Bangkok
  - Investigational Site Number : 764005, Khon Kaen
- United Kingdom (8):
  - Investigational Site Number : 151340, Cambridge, Cambridgeshire
  - Investigational Site Number : 150303, London, London, City of
  - Investigational Site Number : 152361, Salford, Manchester
  - Investigational Site Number : 150455, Manchester, Missouri
  - Investigational Site Number : 154196, Belfast
  - Investigational Site Number : 152287, Birmingham
  - Investigational Site Number : 151123, London
  - Investigational Site Number : 151646, London
- Investigational Site Number : 154212, Hanoi, Vietnam

REFERENCES:
- [Background] Germain DP, Brand E, Burlina A, Cecchi F, Garman SC, Kempf J, Laney DA, Linhart A, Marodi L, Nicholls K, Ortiz A, Pieruzzi F, Shankar SP, Waldek S, Wanner C, Jovanovic A. Phenotypic characteristics of the p.Asn215Ser (p.N215S) GLA mutation in male and female patients with Fabry disease: A multicenter Fabry Registry study. Mol Genet Genomic Med. 2018 Apr 12;6(4):492-503. doi: 10.1002/mgg3.389. Online ahead of print. PMID 29649853
- [Background] Wilcox WR, Feldt-Rasmussen U, Martins AM, Ortiz A, Lemay RM, Jovanovic A, Germain DP, Varas C, Nicholls K, Weidemann F, Hopkin RJ. Improvement of Fabry Disease-Related Gastrointestinal Symptoms in a Significant Proportion of Female Patients Treated with Agalsidase Beta: Data from the Fabry Registry. JIMD Rep. 2018;38:45-51. doi: 10.1007/8904_2017_28. Epub 2017 May 17. PMID 28510034
- [Background] Hopkin RJ, Cabrera G, Charrow J, Lemay R, Martins AM, Mauer M, Ortiz A, Patel MR, Sims K, Waldek S, Warnock DG, Wilcox WR. Risk factors for severe clinical events in male and female patients with Fabry disease treated with agalsidase beta enzyme replacement therapy: Data from the Fabry Registry. Mol Genet Metab. 2016 Sep;119(1-2):151-9. doi: 10.1016/j.ymgme.2016.06.007. Epub 2016 Jun 13. PMID 27510433
- [Derived] Hopkin RJ, Cabrera GH, Jefferies JL, Yang M, Ponce E, Brand E, Feldt-Rasmussen U, Germain DP, Guffon N, Jovanovic A, Kantola I, Karaa A, Martins AM, Tondel C, Wilcox WR, Yoo HW, Burlina AP, Mauer M. Clinical outcomes among young patients with Fabry disease who initiated agalsidase beta treatment before 30 years of age: An analysis from the Fabry Registry. Mol Genet Metab. 2023 Feb;138(2):106967. doi: 10.1016/j.ymgme.2022.106967. Epub 2022 Nov 30. PMID 36709533
- [Derived] Wanner C, Feldt-Rasmussen U, Ortiz A. Plain language summary of a study looking at heart muscle thickness and kidney function in women with Fabry disease who received agalsidase beta treatment. Future Cardiol. 2022 Sep;18(10):755-763. doi: 10.2217/fca-2022-0047. Epub 2022 Sep 8. PMID 36073247
- [Derived] Ortiz A, Abiose A, Bichet DG, Cabrera G, Charrow J, Germain DP, Hopkin RJ, Jovanovic A, Linhart A, Maruti SS, Mauer M, Oliveira JP, Patel MR, Politei J, Waldek S, Wanner C, Yoo HW, Warnock DG. Time to treatment benefit for adult patients with Fabry disease receiving agalsidase beta: data from the Fabry Registry. J Med Genet. 2016 Jul;53(7):495-502. doi: 10.1136/jmedgenet-2015-103486. Epub 2016 Mar 18. PMID 26993266
- [Derived] Germain DP, Charrow J, Desnick RJ, Guffon N, Kempf J, Lachmann RH, Lemay R, Linthorst GE, Packman S, Scott CR, Waldek S, Warnock DG, Weinreb NJ, Wilcox WR. Ten-year outcome of enzyme replacement therapy with agalsidase beta in patients with Fabry disease. J Med Genet. 2015 May;52(5):353-8. doi: 10.1136/jmedgenet-2014-102797. Epub 2015 Mar 20. PMID 25795794